CLINICAL TRIAL: NCT05483010
Title: Pilot Study of Statins in Patients With Clonal Cytopenia of Undetermined Significance (CCUS) and Myelodysplastic Syndromes (MDS)
Brief Title: Statins in Patients With Clonal Cytopenia of Undetermined Significance (CCUS) and Myelodysplastic Syndromes (MDS)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202211020
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Clonal Cytopenia of Undetermined Significance; Myelodysplastic Syndromes
Keywords: CCUS; MDS; Statins; Inflammation
MeSH Terms: conditions — Myelodysplastic Syndromes; Inflammation | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atorvastatin (Experimental): * Choice of statin is at the discretion of the treating physician and may depend on insurance approval.
  * Atorvastatin dosing starts at 80 mg once daily.
  * In the absence of disease progression or intolerable side effects, patients may receive up to 12 months of treatment.
  * If a patient switches statins due to toxicity, treatment time is still limited to 12 months total (ie, if a patient receives 6 months of atorvastatin and switches to rosuvastatin, the duration of rosuvastatin will be no more than 6 months).
  Interventions: Drug: Atorvastatin
- Rosuvastatin (Experimental): * Choice of statin is at the discretion of the treating physician and may depend on insurance approval.
  * Rosuvastatin dosing starts at 40 mg once daily.
  * In the absence of disease progression or intolerable side effects, patients may receive up to 12 months of treatment.
  * If a patient switches statins due to toxicity, treatment time is still limited to 12 months total (ie, if a patient receives 6 months of atorvastatin and switches to rosuvastatin, the duration of rosuvastatin will be no more than 6 months).
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin is commercially available.
  Other Names: Lipitor
  Arms: Atorvastatin
Drug: Rosuvastatin — Rosuvastatin is commercially available.
  Other Names: Crestor
  Arms: Rosuvastatin

SUMMARY:
Patients with clonal cytopenia of undetermined significance (CCUS) and lower-risk myelodysplastic syndromes (MDS) have a life expectancy of 5 to 10 years. Mortality in these patients results from progression of disease to higher-risk MDS or acute myeloid leukemia (AML) and cardiovascular events. Currently there are no FDA-approved treatments with the potential to improve survival of patients with CCUS and lower-risk MDS. Statins are an appealing class of drugs to consider in this situation as preclinical data support their potential to suppress progression of myeloid malignancy, and they have a well-established role in prevention of major cardiovascular events. This is a pilot study to explore the role of statins in treatment of patients with CCUS and lower-risk MDS. In this study, change in inflammatory biomarkers and variant allele frequency (VAF) of somatic mutations will be used as a surrogate marker of response to statin therapy. The hypothesis is that the use of statins at diagnosis of CCUS or lower-risk MDS will reduce inflammation and delay or prevent the expected increase in the VAF of somatic mutations over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CCUS or lower-risk MDS as defined below:

  * CCUS is defined as the presence of somatic mutation(s) in recurrently mutated genes identified through the clinical MyeloSeq assay with a VAF ≥ 2% in the absence of bone marrow morphology/cytogenetic changes diagnostic of MDS PLUS unexplained persistent cytopenia in at least one lineage for at least 6 months:

    * Hemoglobin < 11.3 g/dL in females or < 13 g/dL in males
    * ANC < 1.8 x 109/L
    * Platelets < 150 x 109/L
  * MDS is defined using the WHO 2016 definition and classified into lower-risk if IPSS-R score is ≤ 3.5 . Lower-risk MDS will be required to have at least one mutation in a recurrent mutated gene with a VAF ≥ 2%.
* Patient must be transfusion independent.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* CCUS patients with cytogenetic change alone.
* Current or prior use of disease-modifying therapy (e.g., lenalidomide, Luspatercept, Imitelstat, HMAs, venetoclax) with any dose within the last 3 months, with the exception of concurrent use of erythropoetin stimulating agents
* Prior use of a statin within 1 year prior to start of treatment.
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence active of disease.
* Currently receiving any investigational agent for CCUS/MDS. The minimum interval between the last dose of investigational agent used for CCUS/MDS and Day 1 of this trial should be 5 half-lives of the investigational agent.
* A history of allergic reactions or intolerance attributed to compounds of similar chemical or biologic composition to atorvastatin, rosuvastatin, any other statin, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic infection, sepsis, or active liver disease (acute liver failure, decompensated cirrhosis, or persistent elevation in ALT or AST > 3 x ULN), or any other comorbidity that would preclude statin use based on FDA recommendation.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Patients with HIV and HCV are not eligible for the trial if they are concomitantly receiving active treatment for HIV/HCV given the concern for potential drug interactions. The minimum interval between the last dose of antiviral and enrollment into the study should be 28 days or 5 half-lives of the antiviral drug, whichever is longer. The liver function profile of eligible HIV/HCV patients must be within the acceptable limits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in hs-CTRP levels in peripheral blood during statin therapy | Pre-treatment, every 3 months while on treatment, end of treatment, 3 months after end of treatment and time of progression (estimated to be 15 months)

SECONDARY OUTCOMES:
Change in allele burden (VAF) of somatic mutation | Pre-treatment, every 3 months while on treatment, end of treatment, 3 months after end of treatment and time of progression (estimated to be 15 months)
  -Assessed by next generation sequencing (NGS) performed on peripheral blood/bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Amber Afzal, M.D., MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Washington University in St Louis supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required (as a condition of research awards and/or as otherwise required).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication.
Access Criteria: Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu